CLINICAL TRIAL: NCT04340713
Title: Construction and Evaluation of Supportive Care for Patients With Prostate Cancer During Hormonal Therapy
Brief Title: The Effect of Information Support Program on Self-efficacy of Prostate Cancer Patients During Hormonal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhenqi Lu, Director of Nusing Administration, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 1805185-14
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Information Support
Keywords: Prostate cancer; hormonal therapy; information support
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information support group (Experimental): The experimental group was given information support program intervention on the basis of routine information communication.
  Interventions: Other: information support program
- Routine care group (No Intervention): The control group was given routine information communication.

INTERVENTIONS:
Other: information support program — According to the established information support program for prostate cancer patients during hormonal therapy, information support and guidance on disease knowledge, symptom management, life care and other aspects are provided to patients through face-to-face communication, telephone, written information, network and other ways.
  Arms: Information support group

SUMMARY:
The incidence rate of prostate cancer has been increasing rapidly in China in recent years. However, a large number of studies have shown that, patients with prostate cancer during hormonal therapy generally face the imbalance of high information demand and low information acquisition, which affects their mental health and quality of life, and even reduces their treatment adherence. Thus, the investigators designed a randomized control study in one cancer center in Shanghai. Prostate cancer patients during hormonal therapy were followed up in the urology clinic and ward, and then they were randomly divided into control group and experimental group according to the order of enrollment. The control group was given routine information communication, and the experimental group was given information support program intervention on this basis. The effects of the intervention was evaluated after 3 months. The investigators expected that the information support program would be helpful to improve patients' self-efficacy level, and to enhance their confidence in self-management and coping with difficulties, so as to improve patients' adherence of health behaviors and improve their health-related quality of life.

DETAILED DESCRIPTION:
The incidence rate of prostate cancer has been increasing rapidly in China in recent years. It has gradually become one of the most common malignant tumors of the urinary system in men. However, a large number of studies have shown that, patients with prostate cancer during hormonal therapy generally face the imbalance of high information demand and low information acquisition, which affects their mental health and quality of life, and even reduces their treatment adherence. Thus, the investigators designed a randomized control study in one cancer center in Shanghai. Prostate cancer patients during hormonal therapy were followed up in the urology clinic and ward of a cancer center in Shanghai from July to October 2019 ,then patients were randomly divided into control group and experimental group according to the order of enrollment. The control group was given routine information communication, and the experimental group was given information support program intervention on this basis. The effects of the intervention was evaluated after 3 months. The investigators expected that the information support program would be helpful to improve patients' self-efficacy level, and to enhance their confidence in self-management and coping with difficulties, so as to improve patients' adherence of health behaviors and improve their health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

Patients were diagnosed as prostate cancer by biopsy or operation; At the initial stage of hormonal therapy for prostate cancer (0-3 months); The time of hormonal therapy was expected more than 6 months; Master basic operation skills of the app "wechat", or can simply use it after learning; Primary school education or above; Age < 80; Have a clear sense of reading, understanding and communication skills; Willing to participate in this study and sign informed consent.

Exclusion Criteria:

Have received castration operation; Combined with other tumors; Combined with other serious endocrine diseases; Serious diseases in heart, brain, lung or other important organs.

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Information satisfaction | 3 months
  EORTC QLQ-INFO25, a questionnaire include 25 items was used to measure patients' information acquisition and information satisfaction on disease, medical tests, treatments, and other aspects.
Self-efficacy | 3 months
  SUPPH, the Chinese version include 28 items was used to measure patients' level of self-efficacy and confidence in coping.

SECONDARY OUTCOMES:
Mastery of disease knowledge | 3 months
  A self-designed questionnaire covering a total of 18 items was used to measure patients' knowledge on prostate cancer, review, hormonal therapy, and healthy life style.
Adherence of healthy behaviors | 3 months
  A self-designed questionnaire covering a total of 10 items was used to measure patients' adherence of healthy behaviors on the aspects of bad habits, diet, physical exercise, medication, and reviews.
Health-related quality of life | 3 months
  AMS, a questionnaire include 17 items was used to measure patients' somatic symptom, psychological symptom, sexual symptom, and patients' health-related quality of life.
the serum PSA level | 3 months
  The serum PSA (prostate cancer specific antigen) level was recorded at baseline and 3 months after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Rui Yang, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided